CLINICAL TRIAL: NCT00448175
Title: Overactive Bladder Innovative Therapy Trial
Brief Title: Overactive Bladder Innovative Therapy Trial (OrBIT)
Acronym: OrBIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Uroplasty, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPC032006
Record Dates: First submitted 2007-03-15; First posted 2007-03-16 (Estimated); Results first posted 2013-05-16 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-04

CONDITIONS: Overactive Bladder
Keywords: OAB symptoms of urgency, frequency, and urge incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge | interventions — Tolterodine Tartrate

ARMS (1):
- Urgent PC treatment arm (Experimental)
  Interventions: Device: Urgent PC Neuromodulation System; Drug: Tolterodine

INTERVENTIONS:
Device: Urgent PC Neuromodulation System — The Urgent PC Neuromodulation System is a minimally invasive neuromodulation system designed to deliver retrograde access to the sacral nerve through percutaneous electrical stimulation of the tibial nerve. The method of treatment is referred to as Percutaneous Tibial Nerve Stimulation (PTNS).
Drug: Tolterodine

SUMMARY:
The purpose of this study is to compare percutaneous tibial nerve stimulation (PTNS) to drug therapy for the treatment of symptoms of overactive bladder (OAB).

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age
* Experiences OAB with a voiding frequency of at least 8 times per day
* Is ambulatory and able to use a toilet independently and without difficulty

Exclusion Criteria:

* On OAB pharmacotherapy within the previous month
* Primary complaint is stress urinary incontinence
* Has pacemaker or implantable defibrillator
* Has history of heart problems
* Has nerve damage or neuropathy
* Has gastric or urinary retention
* Has uncontrolled narrow-angle glaucoma
* Has known sensitivity to drug ingredients
* Is pregnant or planning to become pregnant during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-06; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan O'Toole, Study Director — Uroplasty, Inc
Locations (1):
- Uroplasty, Inc, Minnetonka, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited by investigator sites with limited advertising
Pre-assignment Details: After 12 weekly PTNS treatments, 35 patients were considered responders (reporting of "Moderately" or "Markedly" improved on the Global Response Assessment (GRA))and allowed to continue in the trial through 12 months.
Groups:
- Urgent PC Treatment Arm: The Urgent PC Neuromodulation System is a minimally invasive neuromodulation system designed to deliver retrograde access to the sacral nerve through percutaneous electrical stimulation of the tibial nerve. The method of treatment is referred to as Percutaneous Tibial Nerve Stimulation (PTNS).
- 4mg Daily Tolterodine: 90 day prescription for 4mg daily extended-release tolterodine tartrate (Detrol LA)
Period: 12 Weeks PTNS vs. Drug
Arm/Group | Urgent PC Treatment Arm | 4mg Daily Tolterodine
Started | 50 | 50
Completed | 41 | 43
Not Completed | 9 | 7
Period: Continued PTNS Through 12 Months
Arm/Group | Urgent PC Treatment Arm | 4mg Daily Tolterodine
Started | 35 | 0
Completed | 25 | 0
Not Completed | 10 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Urgent PC Treatment Arm | 4mg Daily Tolterodine | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 35 | 68
  >=65 years | 17 | 15 | 32
Age Continuous [Mean (Standard Deviation); unit: years] | 57.5 (15.2) | 58.2 (11.3) | 57.85 (13.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 46 | 94
  Male | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Voids at 12 Weeks
Description: To demonstrate that the Urgent PC system is as effective as or more effective (noninferior) than tolterodine (Detrol LA) in changing the frequency of urinary voids per day after 12 weeks of therapy. The voiding diaries completed at 12 weeks were compared to the baseline voiding diaries.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: Voids/day
Arm/Group | Urgent PC Treatment Arm | 4mg Daily Tolterodine
Number analyzed (Participants) | 41 | 43
Voids/day | -2.4 (4) | -2.5 (3.9)

2. Secondary Outcome: Urge Incontinence Episodes at 12 Weeks
Time Frame: 12 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Volume Voided at 12 Weeks
Time Frame: 12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: OAB Quality of Life at 12 Weeks
Time Frame: 12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Known Side Effects Through 12 Weeks
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Urgent PC Treatment Arm | 4mg Daily Tolterodine
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 6/50 | 4/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Urgent PC Treatment Arm (N=50) | 4mg Daily Tolterodine (N=50)
Bruising (Surgical and medical procedures) | 1 (3) | 0 (0)
Leg cramp (Surgical and medical procedures) | 2 (2) | 0 (0)
Redness/Inflammation at needle site (Surgical and medical procedures) | 1 (2) | 0 (0)
Pressure/discomfort at needle site (Surgical and medical procedures) | 3 (3) | 0 (0)
Vasovagal response to needle placement (Surgical and medical procedures) | 1 (1) | 0 (0)
Jolt felt in leg during treatment (Surgical and medical procedures) | 1 (1) | 0 (0)
Blurred Vision (Surgical and medical procedures) | 0 (0) | 1 (2)
Headache (Surgical and medical procedures) | 0 (0) | 1 (1)
Constipation (Surgical and medical procedures) | 0 (0) | 1 (1)
Increase urgency/frequency (Surgical and medical procedures) | 0 (0) | 1 (1)
Severe Dizziness (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No